CLINICAL TRIAL: NCT03372642
Title: Valutazione Dell'Efficacia Dell'Endortesi Senotarsica Nella Correzione Della Sindrome Pronatoria Nel Bambino (Flatfoot)
Brief Title: Effectiveness of Subtalar Arthroereisis With Endorthesis for Pediatric Flexible Flat Foot
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: EndSP
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Flatfoot; Pediatric ALL
MeSH Terms: conditions — Flatfoot; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subtalar endorthesis: Patients who underwent subtalar endorthesis for flexible pediatric flatfoot
  Interventions: Device: Subtalar endorthesis

INTERVENTIONS:
Device: Subtalar endorthesis — Subtalar arthroereisis with endorthesis for pediatric flexible flat foot

SUMMARY:
Pediatric flexible flatfoot is sometimes asymptomatic but it can also cause physical impairment, pain, and difficulty walking. We evaluate the radiographic effectiveness of intervention of subtalar arthroereisis with endorthesis for pediatric flexible flatfoot with final follow-up at skeletal maturity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* age ≥ 14 years at the time of the visit
* patients who underwent subtalar endothesis for the treatment of the pediatric flexible flatfoot from January 2011 to March 2015.

Exclusion Criteria:

* age <14 years at the time of the visit
* patients with comorbidities that make it difficult to return to the hospital for consultation or who have removed the device for discomfort
* female patients who do not exclude (by self-declaration, as clinical practice) a state of pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively review 60 consecutive patients who underwent surgical treatment with subtalar arthroereisis for pediatric flexible flatfoot at the authors' institution from January 2011 to March 2015.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
lateral talocalcaneal angle | 1 day
  lateral talocalcaneal angle (LTC) on the lateral view of the radiographs: it is traced between the long axis of the talus and the plantar surface of the calcaneus

SECONDARY OUTCOMES:
AOFAS | 1 day
  American Orthopaedic Foot & Ankle Society (AOFAS) ankle-hindfoot scale. It is a measure of ankle and hidfoot function. It comprises nine questions and covers three categories: pain (40 points), function (50 points) and alignment (10 points). These are all summed together for a maximun score of 100 points (best otucome) and a minimum score of 0 (worst outcome). It includes a mixture of questions that are both subjective and objective in nature.
SEFAS | 1 day
  Self-reported foot and ankle score (SEFAS)
SF-12 | 1 day
  12-Item Short Form Health Survey (SF-12) with its Mental and Physical Component Scores (MCS and PCS)
Meary's angle | 1 day
  Meary's angle (MA) on the lateral view of the radiographs, also known as talar-first metatarsal angle: it is formed by a line through the long axis of the talus and the axis of the first metatarsal (the negative values indicate a plantar apex of the angle as it happens in the flatfeet
Calcaneal pitch angle | 1 day
  Calcaneal pitch angle on the lateral view of the radiographs: it is subtended by the intersection of a line parallel to the floor with a line connecting the two most inferior points on the calcaneus
Anteroposterior talonavicular coverage angle | 1 day
  Anteroposterior talonavicular coverage angle (APTN) on the anteroposterior view of the radiographs: it is the angle between the lines connecting the endpoints of the talar and navicular articular surfaces
Talonavicular uncoverage percent | 1 day
  Talonavicular uncoverage percent (TNU) on the anteroposterior view of the radiographs: it is a ratio between the angle subtended by the line connecting the endpoints of the talar articular surface and a line drawn from the midpoint of the previous line and the medial endpoint of the navicular articular surface. It indicates the percentage of the talar head not covered by the navicular